CLINICAL TRIAL: NCT00067392
Title: Prospective Evaluation of Immediate Temporized Implants
Brief Title: Evaluation of Implants Placed Immediately or Delayed Into Extraction Sites
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Implant Innovations (Industry)
Responsible Party: Michael S Block, LSU School of Dentistry
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: NIDCR-14185; R01DE014185 (NIH)
Record Dates: First submitted 2003-08-15; First posted 2003-08-20 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2008-07

CONDITIONS: Dental Caries
Keywords: Partial edentulism; Bone atrophy; Bone healing
MeSH Terms: conditions — Dental Caries | interventions — Dental Implants

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Procedure: Dental Implant — Dental Implant 4 month time frame

SUMMARY:
The purpose of this study is to determine the difference in success when placing implants immediately into an extraction site compared to delaying the implant placement until the extraction site has healed. In addition, the level of bone around the implants will be compared to determine if one method leads to better results over time.

DETAILED DESCRIPTION:
This revised application is a clinical trial designed to evaluate crestal bone level changes when implants are placed into extraction sites and immediately provisionalized. Extraction of maxillary incisor teeth is a common procedure as documented in our school clinics. Traditional treatment when a tooth is extracted includes a period of healing followed by placement of an implant. Our preliminary data indicates that the delayed approach results in labial bone loss with resultant horizontal deficiency in over 50% of cases, requiring hard and soft tissue grafting to achieve a functional result. Additional preliminary data indicates that grafting the extraction site and/or immediate implant placement and provisionalization results in a functional restoration, without the need for additional adjunctive grafting procedures. It is unclear how the crestal bone levels change during healing of the extraction site prior to implant placement, in contrast to immediate implant placement, with immediate provisionalization with a crown. We hypothesize that there will be differences in the crestal bone levels (primary endpoint), and differences in soft tissue levels and indices (secondary endpoints) between implants immediately temporized, placed either delayed or immediately after tooth extraction, with more bone loss in the immediate placement group (experimental) compared to the delayed placement group (control). The long-term goal is to determine if the crestal bone remodeling after tooth extraction or the apical position of the implant determines the final level of the crestal bone. Two groups of 45 patients will be evaluated. All subjects will have a single rooted maxillary tooth extracted. One group will have the socket grafted with mineralized bone and allowed four months prior to implant placement. The crestal bone in this group will have remodeled during the four months of healing prior to implant placement. The second group will have the implant placed immediately after tooth extraction, thus the crestal bone will remodel in the presence of the implant and the immediately placed temporary restoration, as a one-stage procedure. For both groups, the implants will be immediately temporized with a crown after implant placement. Standardized hard and soft tissue data will be collected pre-extraction as baseline, and then prospectively for at least two years in this trial, to compare the methods and contrast the effectiveness of the proposed immediate restoration therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be willing to be present for examination two times a year for at least three years, as well as maintenance cleanings twice a year 3 months prior to the data collection visit.
* All patients will be free of uncontrolled diabetes (any type), existing malignancy, and will not be receiving any therapy that suppresses their immune system, such as radiation, chemotherapy, or chronic steroid usage
* Need for extraction of a single rooted maxillary central or lateral incisor, canine, or premolar, with no signs of acute infection (purulent exudate, erythema, pain, and swelling).
* Patients will have bone present on all surfaces of the tooth within 3 mm of the gingival margin of the planned restoration, in order to provide sufficient bone to circumferentially cover the implant.
* All patients will have adequate space for satisfactory restoration of the edentulous space.
* Each patient's dentition will be free of active periodontal disease or exhibit controllable periodontal disease such that their teeth will clinically be non-mobile and have probing depths less than 3 mm.
* All prospective sites will have at least 2mm of attached or keratinized gingiva.
* The crestal bone width should be enough to accommodate either a 3.75 diameter implant for the central incisor, canine, and premolar sites, or a 3.25 mm diameter implant for the lateral incisor tooth sites. Bone height should be at least 14 mm for accommodation of the implant.

Exclusion Criteria:

* Patients with labial dehiscence defects greater than 3 mm from the proposed gingival margin of the planned restoration will be excluded from this study.
* Patients who cannot come for follow up due to conflicts of schedules will not be accepted into the study.
* Patients with advanced cardiovascular, pulmonary, renal, liver disease that place them in an ASA III or IV rating will be excluded. Post-menopausal women with known osteoporosis as determined by their medical internist, will be excluded. Patients with known alcohol abuse will be excluded.

Ages: 21 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2003-11; Primary Completion 2008-04 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Crestal bone levels adjacent to the implants | 4 months

SECONDARY OUTCOMES:
Position of the papillary complex and facial gingival margin, and indicator of the inflammatory state of the perimplant tissues. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Block, DMD, Ph.D, Principal Investigator — LSU School of Dentistry
Locations (1):
- LSU School of Dentistry, New Orleans, Louisiana, United States